CLINICAL TRIAL: NCT00116792
Title: PROVIDENCE: Prevention of Restenosis With Oral Rosiglitazone and the Vision Stent in Diabetics With de Novo Coronary Lesions
Brief Title: PROVIDENCE:Prevention of Restenosis With Oral Rosiglitazone and the Vision Stent in Diabetics With Coronary Lesions
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gold, Herman K., MD (Individual)
Collaborators: Guidant Corporation (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 2003P-001717
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
Keywords: CAD; Diabetes Mellitus; Restenosis; ppar gamma; glitazone
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus | interventions — Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention (PCI)

SUMMARY:
We hypothesize that the combination of the thin-strut MULTI-LINK (i.e. VISION(tm) and/or MINI-VISION(tm)) stent and pharmacologic therapy with the oral PPAR-gamma agonist rosiglitazone will significantly reduce restenosis after intracoronary stenting in type 2 diabetic patients. This approach would present a more effective and economical alternative to the use of drug-eluting stents to reduce stent restenosis.

ELIGIBILITY:
Inclusion Criteria:

* The patients must be >18 years of age;
* Patients must be previously diagnosed with type 2 diabetes with documented treatment with insulin, oral hypoglycemics, or diet controlled by medical history. (Undocumented or newly diagnosed diabetics must fulfill the American Diabetes Association Criteria-Report of the Expert Committee on the Diagnosis and Classification of Diabetes Mellitus (Diabetes Care 2003;26:S5-20)).
* Diagnosis of angina pectoris defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II-III) OR patients with documented silent ischemia;
* Treatment of lesions in native coronary arteries requiring stenting. A total of two separate lesions can be stented, located either in the same vessel (at least 10 mm or 1 cm apart) or in two separate vessels. Additional stents may be used for procedural complications such as dissections.
* Patient is willing to comply with the specified follow-up evaluation;
* Patient must provide written informed consent prior to the procedure using a form that is approved by the local Institutional Review Board.
* Target lesion is ≥2.0 mm to ≤3.5mm in diameter (visual estimate);
* Individual lesions are ≤25 mm in length located in a native coronary artery;
* Target lesions are de novo lesions in native coronary vessels;
* Target lesion stenosis is ≥50% and <100% (visual estimate);

Exclusion Criteria:

* Patient has experienced an ST-segment elevation myocardial infarction within the preceding 24 hours.
* Ejection fraction ≤40%; class III-IV CHF
* Active liver disease (ALT>2.5 times upper limit of normal)
* Woman of child-bearing potential unless demonstrated 1) negative pregnancy test and 2) clear intention of an accepted method of contraception for eight months after enrollment
* Totally occluded vessel (TIMI 0 grade flow);
* Impaired renal function (creatinine ≥2.5 mg/dL);
* Target lesion involves bifurcation including a side branch ≥2.5 mm in diameter (either stenosis of both main vessel and major branch or stenosis of just major branch) that would require side branch stenting which is likely to occur if side branch is diseased and intended to be stented;
* Previous brachytherapy of target vessel;
* Recipient of heart transplant;
* Patient with a life expectancy less than 12 months;
* Known allergies to cobalt, chromium, nickel, aspirin, clopidogrel bisulfate (Plavix®) and/or ticlopidine (Ticlid®), heparin, and/or rosiglitazone (Avandia®), that cannot be medically managed;
* Any significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study;
* Currently participating in an investigational drug or another device study;
* Any contraindication to glycoprotein IIb/IIIa inhibitor therapy;
* Current use of any TZD, i.e. rosiglitazone (Avandia®) or pioglitazone (Actos®)
* Chronic or relapse/remitting hemolytic condition
* Unprotected left main coronary disease with >50% stenosis;
* Patients admitted for treatment of diabetic ketoacidosis >2 times in the past six months (brittle diabetics) and/or the suspicion of type I diabetes;
* Target lesion is in a saphenous venous graft or internal mammary graft;
* Target lesion is due to restenosis
* 3 vessel coronary artery disease defined as ≥70% ischemia producing lesions in 3 different epicardial coronary arteries all requiring revascularization (i.e. main left main equivalent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2004-03

PRIMARY OUTCOMES:
In-stent and In-segment late lumen loss

SECONDARY OUTCOMES:
In-stent mean percent diameter stenosis (%DS) and binary restenosis as measured by QCA at post-procedure and at 8 months
TLR and TVR at 30 days, and 8 months post procedure
TVF defined as cardiac death, MI, or TVR at 30 days, 8 months and l year post-procedure
Composite of Major Adverse Cardiac Events (MACE)
The association of metabolic factors and inflammatory indices including glycemia (HgbA1C), diabetic therapy other than TZDs, HSCRP, coagulation (PAI-1, FIB) and inflammatory marker levels (ADI, MPO, &MMP-9) with the risk for restenosis
Target HgbA1C≤7 for all patients enrolled
Coronary artery stenosis progression in at least one non-stented lesion
Coronary artery stenosis regression in at least one non-stented lesion
Culprit (i.e. stented artery) artery stenosis progression/regression by intravascular ultrasound (IVUS)
(There are 3 more secondary endpoints not listed here.)

CONTACTS AND LOCATIONS:
Overall Officials: Herman K Gold, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States